CLINICAL TRIAL: NCT03386240
Title: Antibacterial-coated Sutures at Time of Cesarean
Acronym: ASTC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-0305
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Surgical Site Infection; Surgical Wound Infection; Cesarean Section; Infection; Cesarean Section Complications
MeSH Terms: conditions — Surgical Wound Infection; Infections | interventions — Population Groups; Polyglactin 910; glycolide E-caprolactone copolymer; Triclosan; Control Groups

STUDY DESIGN:
Intervention Model Description: Double-blinded controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: A confidential computer-generated simple randomization scheme will be prepared and provided on an ongoing basis. A randomization log will be used to track the randomization process. Patients will be masked to the suture material. Both suture types look similar. Patient, surgeons, and staff ascertaining the outcomes will be masked for the suture type.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vicryl-plus, monocryl-plus, PDS-plus (Triclosan-coated Sutures (Experimental): Use of Monocryl Plus, Vicryl Plus and PDS Plus Suture (Triclosan-coated sutures) will be used exclusively throughout the entire procedure.
  Interventions: Drug: Vicryl-plus, monocryl-plus, PDS-plus (Triclosan-coated Sutures)
- Vicryl, monocryl, PDS (not coated with triclosan) (Placebo Comparator): Use of Monocryl, Vicryl and PDS Suture (equivalent uncoated sutures) will be used exclusively throughout the whole procedure.
  Interventions: Other: Vicryl, monocryl, PDS (not coated with triclosan)

INTERVENTIONS:
Drug: Vicryl-plus, monocryl-plus, PDS-plus (Triclosan-coated Sutures) — The intervention consists of using Plus group (Triclosan-coated Sutures)
  Other Names: Plus group
  Arms: Vicryl-plus, monocryl-plus, PDS-plus (Triclosan-coated Sutures
Other: Vicryl, monocryl, PDS (not coated with triclosan) — Consists of equivalent sutures (not coated with triclosan) during cesarean delivery.
  Other Names: Control group
  Arms: Vicryl, monocryl, PDS (not coated with triclosan)

SUMMARY:
Abdominal closure with antibacterial-coated sutures has been shown to reduce wound infections after a number of surgical procedures, but none of the previous trials included cesarean delivery. Our objective is to determine whether use of antibacterial-coated sutures reduces surgical site infection (SSI) after cesarean delivery.

DETAILED DESCRIPTION:
A review of 18 studies demonstrated a significant benefit of antimicrobial coated sutures in reducing SSI (RCTs: OR 0.72; 95% CI 0.59-0.88; observational studies: OR 0.58; 95% CI 0.40-0.83). As there are no clinical trials focusing on cesarean delivery, and because the risk factors and pathogenesis for post-cesarean SSI may not mirror other procedures, further data is needed before generalizing the WHO recommendations to cesarean procedures.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age.
* Women ≥ 24 weeks' viable gestation.
* To undergo cesarean delivery.

Exclusion Criteria:

* Patient unwilling or unable to provide consent.
* No prenatal care or a non-resident patient who is unlikely to be followed-up after delivery.
* Immunosuppressed patients: i.e., taking systemic immunosuppressant or steroids (e.g. transplant patients; not including steroids for lung maturity), HIV with CD4<200, or other.
* Decision to use other than suture closure (e.g. secondary wound closure, mesh closure).
* Skin infection.
* Coagulopathy.
* High likelihood of additional surgical procedure beyond cesarean (e.g. scheduled hysterectomy, bowel or adnexal surgery).
* Allergy to Triclosan.
* Incarcerated individuals.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female admitted to labor and delivery
Enrollment: 1122 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Composite of endometritis and/or wound infection and/or other post-cesarean infections | occurring within 30 days of delivery
  surgical site infection after cesarean

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Bush, M.D., Principal Investigator — University of Texas Medical Branch in Galveston
Locations (1):
- University of Texas Medical Branch in Galveston, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No